CLINICAL TRIAL: NCT03034408
Title: Effects of Nalmefene and Baclofen on Impulsivity in Subjects With Alcohol Use Disorder and Healthy Control Subjects: A Randomized, Placebo-controlled Study
Brief Title: Nalmefene, Baclofen and Impulsivity in Subjects With Alcohol Use Disorder and Healthy Control Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Daniele Zullino (Other)
Responsible Party: Sponsor-Investigator, Prof. Daniele Zullino, Prof., University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-00160
Record Dates: First submitted 2016-11-03; First posted 2017-01-27 (Estimated); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Alcohol Use Disorder
Keywords: Impulsivity; Nalmefene; Baclofen
MeSH Terms: conditions — Alcoholism; Impulsive Behavior | interventions — nalmefene; Baclofen; Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alcohol Use Disorder (Other): 30 patients with DSM-5 Diagnosis of Alcohol Use Disorder, at least moderate (303.90/F10.20) : Nalmefene 18mg, Baclofen 10mg, Placebo Oral Capsule
  Interventions: Drug: Nalmefene; Drug: Baclofen; Drug: Placebo Oral Capsule
- Healthy Control (Other): 30 sex and age-matched healthy controls : Nalmefene 18mg, Baclofen 10mg, Placebo Oral Capsule
  Interventions: Drug: Nalmefene; Drug: Baclofen; Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Nalmefene
  Other Names: Selincro
Drug: Baclofen
  Other Names: Lioresal
Drug: Placebo Oral Capsule
  Other Names: Mannitol

SUMMARY:
Impulsivity is a central feature of addiction. Nalmefen is an authorized treatment for alcohol addiction. Baclofen has empathically been advocated to have some efficacy in this indication. The aim of the present study is to test the effect of Nalmefene and Baclofen on impulsivity.

Primary study objective: To examine the effect of Nalmefene and Baclofen on impulsivity (as measured by the Stop Signal Task) in subjects with alcohol use disorder and healthy control subjects.

Main secondary study objectives: To examine the effect of Nalmefene and Baclofen on risk taking (as measured by the Balloon Analogue Risk Task) and on the preference for small immediate rewards over large delayed rewards (as measured by the Delay Discounting Task). To compare subjects with alcohol use disorder and healthy control subjects on these tasks.

Primary study outcome: Stop-signal reaction time in the Stop-Signal Task Main secondary study outcomes: Equivalence point in the Delay-Discounting Task and Average number of pumps delivered in the Balloon Analogue Risk Task

Study Design: Randomized, placebo control, cross-over, single-dose

ELIGIBILITY:
Inclusion Criteria:

* 30 patients with DSM-5 Diagnosis of Alcohol Use Disorder, at least moderate (303.90/F10.20),
* 30 sex and age-matched healthy controls,
* over 18, informed consent.

Exclusion Criteria:

* opiate-treatment,
* contra-indications for Nalmefene and/or Baclofen,
* unstable psychiatric disorder,
* pregnancy,
* acute withdrawal syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-07-01; Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Change in "Stop-signal reaction time" in the Stop-Signal Task | 0 and 2 hours post-dose
  Before-drug/after-drug difference of the stop-signal reaction time in the Stop Signal Task at Visit 2, Visit 3 and Visit 4.

SECONDARY OUTCOMES:
Change in "Equivalence point" in the Delay-Discounting Task | 0 and 2 hours post-dose
  Before-drug/after-drug difference of the Equivalence point" in the Delay-Discounting Task at Visit 2, Visit 3 and Visit 4.
Change in "Average number of pumps" delivered in the Balloon Analogue Risk Task | 0 and 2 hours post-dose
  Before-drug/after-drug difference of the "Average number of pumps" delivered in the Balloon Analogue Risk Task at Visit 2, Visit 3 and Visit 4.

CONTACTS AND LOCATIONS:
Overall Officials: Daniele F Zullino, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Service d'Addictologie, Hôpitaux Universitaires de Genève, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: website related to the study — http://www.hug-ge.ch/addictologie/recherche